CLINICAL TRIAL: NCT07118059
Title: Effects of Adjunct Omega-3 Long-chain Polyunsaturated Fatty Acids in Pulmonary Tuberculosis Patients: An Early Bactericidal Activity and Inflammatory Activity Trial
Brief Title: Effects of Adjunct Omega-3 Long Chain Polyunsaturated Fatty Acids in Pulmonary Tuberculosis Patient: an Early Bactericidal Activity and Inflammatory Trial
Acronym: TREAT 3
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: North-West University, South Africa (Other)
Collaborators: Perinatal HIV Research Unit of the University of the Witswatersrand (Other)
Responsible Party: Principal Investigator, Linda Malan, Prof, North-West University, South Africa
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TREAT 3; 20250308 (Other: South African Health Products Regulatory Authority); 250209 (Other: University of Witwatersrand Human Research Ethics Committee (medical))
Record Dates: First submitted 2025-08-04; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: Tuberculosis; Inflammation Biomarkers; Liver Function Tests; Iron Status; Metabolomics; Nutritional Status; Clinical Outcomes
Keywords: Pulmonary tuberculosis; Patients; adjunct omega-3 long chain polyunsaturated fatty acid; early bactericidal; safety trial
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Pulmonary | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Intervention Model Description: This is double blinded placebo controlled early bactericidal activity and early inflammatory activity phase two clinical trial. Participants will be randomly assigned to either receive standard of care as per South African National TB guidelines (2014) plus n-3 LCPUFA in the treatment arm or standards of care plus placebo (high linoleic sunflower oil ). The study will be a single trial study done at the Perinatal HIV research Unit in Matlosana
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Omega 3 Long chain Polyunsaturated fatty acid (Experimental): 20 Participant will be in this arm, randomized for sex and HIV status. Participant in the intervention group will receive 3- 1g fish oil capsules capsules to take with their TB treatment of Omega 3 (real thing mega omega supreme). These capsules provide approximately 2g of EPA and DHA
  Interventions: Dietary Supplement: Omega-3 (EPA+DHA)
- High Linoleic sunflower oil (Placebo Comparator): The placebo group will also consist of 20 participant randomized and stratified for sex, HIV status. They will also receive 3 1g capsules of high linoleic sunflower oil that has been encapsulated using the specification and dimension of the omega 3 real thing capsules to closely match the intervention
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Omega-3 (EPA+DHA) — In this study omega-3 will be the real thing mega omega supreme capsule, it will be used as an adjunct therapy with TB treatment in the intensive phase of treatment. Participant will receive x3, 1g capsules which will provide approximately 2g of EPA and DHA
  Arms: Omega 3 Long chain Polyunsaturated fatty acid
Dietary Supplement: Placebo — This group will receive the placebo, which will be 3 x 1g capsules of high linoleic sunflower oil, the sunflower capsules have been encapsulated to match the dimension of the omega 3 supplement. The capsules will also be given as and adjunct to TB treatment of the intensive phase of TB treatment
  Arms: High Linoleic sunflower oil

SUMMARY:
The goal of this randomized controlled trial is to evaluate the early bactericidal activity, early inflammatory response, and safety of omega-3 long chain polyunsaturated fatty acid (n-3 PUFA) supplementation in adult patients (aged 18- 45 years) with newly diagnosed, bacteriologically confirmed drug-sensitive pulmonary tuberculosis.

The main questions it aims to answers are:

* Does adjunct n-3 LCPUFA supplementation reduce the sputum culture time to positivity
* Does it improve inflammatory markers and TB treatment outcomes compared to placebo Researchers will compare daily supplementation with ~2g n-3 LCPUFA (EPA and DHA ) to placebo (high linoleic sunflower oil) to determine effects on bactericidal activity, inflammation, and clinical outcomes.

Participants will:

* Be randomly assigned to receive either n-3 LCPUFA or Placebo daily for 8 weeks with the intensive phase of TB treatment
* Attend clinical visit baseline, and follow up visit mostly weekly for 2 months and then monthly for 4 months of the continuous phase of TB treatment
* Provide blood, sputum and urine samples for biomarkers and metabolomic analysis
* Undergo assessments of iron status, body composition and muscle strength

DETAILED DESCRIPTION:
Anti-inflammatory omega-3 long-chain polyunsaturated fatty acids (n-3 LCPUFA) supplementation results in improvement of infectious respiratory conditions, yet little evidence in patients with pulmonary tuberculosis (TB) exists. Animal studies have shown that adjunct n-3 LCPUFA optimized treatment outcomes by resolving inflammation, improving immune response, and mitigating iron deficiency and anaemia of inflammation.

This randomized controlled early bactericidal activity (EBA), early inflammatory activity (EIA), and safety trial among patients with newly bacteriologically confirmed adult drug-sensitive pulmonary TB patients (DS-TB), aged 18 - 45 years (n = 40), will investigate the clinical and anti-inflammatory effects of n-3 LCPUFA adjunct treatment for two months.

Patients presenting at Tshepong Hospital, Klerksdorp, North West Province, will receive either ~2 g n-3 LCPUFA (eicosapentaenoic acid (EPA) plus docosahexaenoic acid (DHA)) or placebo (high-linoleic sunflower oil) daily for two months. The primary outcome is sputum culture time to positivity. Secondary outcomes include time to stable culture conversion, proportion of participants converted at 8 weeks, inflammatory markers and safety. Exploratory objectives include iron status, body composition and muscle strength, clinical outcomes, microbial translocation biomarkers, resting energy expenditure, fatty acid composition, plasma lipid mediators, and related metabolomics and gene expression.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 18-45 years
* laboratory confirmed Pulmonary TB defined as a hard copy of a sputum result detected by WHO recommended assay or mycobacteria culture.
* Women of childbearing potential with a negative pregnancy test on enrollment
* All participant irrespective of HIV status who consent to have a HIV test during enrollment.

Exclusion Criteria:

* Comorbid condition with treatment of NSAIDS is indicated
* Institutionalized or incarcerated individuals
* Those on Multiple drug resistance treatment for more than 4 days within the past 6 months or within 1 month to prior to TB treatment initiation
* Pregnant or breastfeeding women or women who become pregnant in the first 4 weeks of the trial will be withdrawn
* show lab safety values: AST or ALT > x3 upper limit of normal (ULN) or Total bilirubin > 2x the ULN, Neutrophils ≤ 700/mm³, Platelets < 50,000/mm³, Haemoglobin < 8 g/dL, Serum creatinine > 2× ULN.
* Are receiving or planning treatment with any of the following in the 3 months before or during the trial:

Anticoagulants Immune-modulating therapy (e.g., cancer treatment, oral/inhaled corticosteroids) Antacids or proton pump inhibitors (PPIs)

* Have a known allergy or sensitivity to fish or fish oil.
* Have a recent history (within 2 years) or current clinical evidence of:

Peptic ulcer disease or GI bleeding Coagulopathy or bleeding disorders Kidney or liver disease requiring hospitalisation Cardiovascular disease or significant risk factors for it

-Are HIV-positive and meet any of the following: CD4 count < 100 cells/mm³ Viral load > 400 copies/mL (if on ART) Not yet on ART but are expected to initiate treatment during the 8-week intervention phase

* Report high-risk alcohol use (average >4 units/day or binge drinking patterns)
* Have any other medical condition or situation that, in the investigator's opinion, may interfere with protocol adherence or data interpretation.
* Plan to relocate from the study area within the next 3 months.
* Are currently using omega-3 or omega-6 supplements and are unwilling to stop for the duration of the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Sputum culture time to positive | TTP will be measured on the following days of the intervention: day 1, day 4, day 7, day 14, day 21, day 30 and day 60
  which is defined as the number of hours between sample inoculation and the detection of microbial growth , A shorter detection time shows that intervention is not working and there is still a higher bacterial load in sputum whilst longer detection time shows improvement in treatment and thus effective intervention

SECONDARY OUTCOMES:
time to stable culture conversion | Sputum cultures to measure time to stable culture conversion will be measured on days: 1,4,7,14,21,30 and 60
  time to stable culture conversion refers to the number of days from the start of TB treatment until a person has two negative sputum cultures with no subsequent positive cultures
Proportion of participants with stable sputum culture conversion | sputum cultures will be collected at day 1, day 4, day 7, day 14, day 21, day 30 and day 60
  Proportion of participants with stable sputum culture conversion, is the number of participant in the group that have two or more negative culture for TB at 8 weeks, if the proportion is more in the omega-3 group compared to placebo than we can conclude that the omega 3 is an effective adjunct therapy.
Safety measures | baseline, day 7, day 30 and day 60
  safety outcomes including the incidence of serious adverse events and abnormal laboratory safety test including; aspartate, aminotransferase, alanine aminotransferase; 3 x the upper limit of normal. Total bilirubin 2x ULN, neutrophil count less than or equal to 700 neutrophils per mm cubed, platelet count less than fifty thousand cells per mm cubed and haemoglobin less than 8g per deciliter and lastly a serum creatinine concentration 2x the upper limit of normal

CONTACTS AND LOCATIONS:
Overall Officials: Linda prof, Principal Investigator — North West University
Locations (1):
- Perinatal HIV research Unit (Matlosana), Klerksdorp, North West, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Time Frame: beginning one year and ending 3 years after publication date
Access Criteria: research who has a methodological sound proposal that has been approved by an independent review committee identified for this purpose

REFERENCES:
- [Background] Hayford FEA, Dolman RC, Ozturk M, Nienaber A, Ricci C, Loots DT, Brombacher F, Blaauw R, Smuts CM, Parihar SP, Malan L. Adjunct n-3 Long-Chain Polyunsaturated Fatty Acid Treatment in Tuberculosis Reduces Inflammation and Improves Anemia of Infection More in C3HeB/FeJ Mice With Low n-3 Fatty Acid Status Than Sufficient n-3 Fatty Acid Status. Front Nutr. 2021 Aug 24;8:695452. doi: 10.3389/fnut.2021.695452. eCollection 2021. PMID 34504860
- [Background] Hayford FEA, Dolman RC, Blaauw R, Nienaber A, Smuts CM, Malan L, Ricci C. The effects of anti-inflammatory agents as host-directed adjunct treatment of tuberculosis in humans: a systematic review and meta-analysis. Respir Res. 2020 Aug 26;21(1):223. doi: 10.1186/s12931-020-01488-9. PMID 32847532
- [Background] Nienaber A, Ozturk M, Dolman RC, Zandberg L, Hayford FE, Brombacher F, Blaauw R, Smuts CM, Parihar SP, Malan L. Beneficial effect of long-chain n-3 polyunsaturated fatty acid supplementation on tuberculosis in mice. Prostaglandins Leukot Essent Fatty Acids. 2021 Jul;170:102304. doi: 10.1016/j.plefa.2021.102304. Epub 2021 May 26. PMID 34082319
- [Background] Nenni V, Nataprawira HM, Yuniati T. Role of combined zinc, vitamin A, and fish oil supplementation in childhood tuberculosis. Southeast Asian J Trop Med Public Health. 2013 Sep;44(5):854-61. PMID 24437320